CLINICAL TRIAL: NCT06565078
Title: Post-marketing Database Survey: a Cohort Study to Evaluate the Safety of Cuvitru in Patients with Primary Immunodeficiency Using the PIDJ2 (Primary Immunodeficiency Database in Japan) Registry
Brief Title: A Database Survey to Evaluate the Safety of Immune Globulin Subcutaneous (Human), 20% Solution in Participants with Primary Immunodeficiency
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: SHP664-403; jRCT2031240293 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-08-20; First posted 2024-08-21 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: Primary immunodeficiency disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Immune Globulin Subcutaneous (Human), 20% Solution: Participants with primary immunodeficiency disease who received Immune Globulin Subcutaneous (Human) 20% infusion in accordance with package insert.
  Interventions: Drug: Immune Globulin Subcutaneous (Human), 20% Solution

INTERVENTIONS:
Drug: Immune Globulin Subcutaneous (Human), 20% Solution — CUVITRU 20% Solution

SUMMARY:
This study is a retrospective database study in Japan to evaluate the safety of Immune Globulin Subcutaneous (Human), 20% Solution in participants with primary immunodeficiency disease (PID). This survey will conduct in use of medical database called PIDJ2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary immunodeficiency (PID) enrolled in the PID patient registry.
2. Participant for whom study drug is entered in the therapeutic drug field on the data set.
3. Participant who is entered the intractable disease diagnosis corresponding to PID in the intractable disease information field.
4. Participant for whom the presence or absence of adverse events has been entered in the column of adverse events.

Exclusion Criteria:

1. Participant for whom study drug has not been entered in the drug name in the medical history field during the period from January 24, 2024 to January 23, 2029.
2. Participant who is not entered the intractable disease diagnosis corresponding to PID in the intractable disease information field.
3. Participant for whom the presence or absence of adverse events has not been entered in the column of adverse events.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience Anaphylactic Reaction as an Adverse Event (AE) | From initial registration in the database or first dose of study drug, whichever came late, up to end date of data period (up to 5 years)
  An AE is defined as any untoward event that occurred in a participant after the first dose of study drug, which does not necessarily have a causal relationship with primary immunodeficiency disease. Number of participants who experience anaphylactic reaction as an AE will be reported.
Number of Participants Who Experience Thromboembolism as an AE | From initial registration in the database or first dose of study drug, whichever came late, up to end date of data period (up to 5 years)
  An AE is defined as any untoward event that occurred in a participant after the first dose of study drug, which does not necessarily have a causal relationship with primary immunodeficiency disease. Number of participants who experience thromboembolism as an AE will be reported.
Number of Participants Who Experience Aseptic Meningitis as an AE | From initial registration in the database or first dose of study drug, whichever came late, up to end date of data period (up to 5 years)
  An AE is defined as any untoward event that occurred in a participant after the first dose of study drug, which does not necessarily have a causal relationship with primary immunodeficiency disease. Number of participants who experience aseptic meningitis as an AE will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/cb1da3ad6f8a4aae??